CLINICAL TRIAL: NCT07390773
Title: Building Relationship, Improving Dialogue, and Growing Empathy (BRIDGE): An Intervention to Support Decision Making for Critically Ill Children
Acronym: BRIDGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00117670; R01HD118955 (NIH)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Decision Making; Neonatal Critical Illness; Pediatric Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the BRIDGE intervention arm, parents will receive a paper-based tool that includes an introduction to decision-making, a values clarification exercise, and a question prompt list. The tool additionally prompts parents to share how they define decision-relevant concepts like quality of life and suffering for their child. The completed tool is shared with the medical team in the electronic health record.
  Interventions: Behavioral: BRIDGE intervention
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: BRIDGE intervention — The BRIDGE intervention includes a paper-based tool that includes an introduction to decision-making, a values clarification exercise, and a question prompt list. The tool additionally prompts parents to share how they define decision-relevant concepts like quality of life and suffering for their child. The completed tool is shared with the health care team in the electronic health record.
  Arms: Intervention

SUMMARY:
Parents of young children in the intensive care unit may be faced with decisions about their child's care. The Building Relationship, Improving Dialogue, and Growing Empathy (BRIDGE) intervention was designed to help support parents as they make decisions for their child and communicate with the health care team. The main questions this study aims to answer are:

1. Do parents who receive the BRIDGE intervention report being better prepared to make decisions for their child?
2. Do parents who receive the BRIDGE intervention report less regret about the decisions they made for their child?

Participants will complete surveys at baseline and approximately 2 weeks, 6 months, and 12 months following enrollment. Some participants will also participate in interviews about their experiences.

ELIGIBILITY:
Inclusion Criteria:

Child inclusion criteria will include:

* Age < 5 years
* Admission to a critical care unit within the preceding 14 days
* An anticipated serious health care decision, defined as a decision about initiating, not initiating, or withdrawing life-sustaining treatment and/or a decision about major intervention.

Parent inclusion criteria will include:

* Age ≥ 18 years
* The ability speak English or Spanish.

Clinician inclusion criteria will include

* Clinical team member of an enrolled child and parent in the intervention group
* Completion of residency or equivalent training.

Exclusion Criteria:

* Children, parents or clinicians who do not meet the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Parent Preparation for Decision Making, as measured by the PrepDM | Approximately 10-14 days following enrollment
  Items can be summed and scored. Score ranges from 0-100, where a higher score indicates higher perceived preparedness for decision making.
Decisional Regret, as measured by the Decision Regret Scale | Approximately 6 and 12 months following enrollment
  Decisional Regret will be measured by the Decision Regret Scale (DRS): The DRS is a 5- item scale used to measure distress or remorse after a health care decision.

SECONDARY OUTCOMES:
Shared Decision Making Quality, as measured by the CollaboRATE (Parent version) | Approximately 10-14 days following enrollment
  This survey is a 3-item measure, and each item can be rated from 0 to 9. Higher scores indicate a higher degree of shared decision making.
Communication Quality, as measured by the Interpersonal Processes of Care (IPC-18) | Baseline; Approximately 10-14 days following enrollment
  For this measure, we will administer the communication and decision making subscales. Each item uses a response scale of 1-5. Higher scores indicate that the labeled interpersonal process occurred more often.
Decisional Conflict, as measured by the Decisional Conflict Scale | Approximately 10-14 days following enrollment; Approximately 6 and 12 months following enrollment
  The Decisional Conflict Scale includes 16 items across 5 domains (score range: 0-100). Higher scores indicate a higher degree of decisional conflict.
Parent Self-efficacy, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions | Approximately 6 and 12 months following enrollment
  Participants will complete the PROMIS self-efficacy for managing chronic conditions measure, which has been adapted for use by parents. This measure assesses parental self-efficacy in managing their child's medications and treatments. Participants will complete the questions in the health care information or decision making domain. Items ask participants to indicate their current level of confidence in each behavior and have 5 response options (range 1-5). Higher scores indicate a higher level of confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Lemmon, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemmon ME, Bansal S, Nanduri N, Davalos A, Glass HC, Lord B, Moline K, Pilon B, Sharpe R, Brandon D, Hong H, Samsa G, Cox CE, Pollak KI. Feasibility of an Intervention to Support Shared Decision-Making for Critically Ill Infants. J Pediatr. 2025 Aug;283:114632. doi: 10.1016/j.jpeds.2025.114632. Epub 2025 May 2. PMID 40319938